CLINICAL TRIAL: NCT03315143
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study to Demonstrate the Effects of Sotagliflozin on Cardiovascular and Renal Events in Patients With Type 2 Diabetes, Cardiovascular Risk Factors and Moderately Impaired Renal Function
Brief Title: Effect of Sotagliflozin on Cardiovascular and Renal Events in Participants With Type 2 Diabetes and Moderate Renal Impairment Who Are at Cardiovascular Risk
Acronym: SCORED
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: study terminated due to business decision
Sponsor: Lexicon Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EFC14875; 2017-002644-32; U1111-1187-8703 (Other: UTN)
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Results first posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-09

CONDITIONS: Heart Failure; Type 2 Diabetes Mellitus; Chronic Kidney Diseases
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sotagliflozin (Experimental): Sotagliflozin 200 mg tablet once daily, with possible up-titration in the first 6 months to 400 mg, for up to 28.9 months.
  Interventions: Drug: Sotagliflozin
- Placebo (Placebo Comparator): Matching placebo to sotagliflozin 200 mg once daily, with possible up-titration in the first 6 months to matching placebo to sotagliflozin 400 mg, for up to 29.6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sotagliflozin — Sotagliflozin was administered as a tablet(s), orally once daily.
  Other Names: SAR439954
  Arms: Sotagliflozin
Drug: Placebo — Placebo was administered as a tablet(s) (identical to the sotagliflozin tablet in appearance), orally once daily.
  Arms: Placebo

SUMMARY:
The primary objective of the study was to compare the effect of sotagliflozin to placebo on total occurrences of cardiovascular (CV) death, hospitalization for heart failure [HHF], and urgent visit for heart failure [HF] in participants with type 2 diabetes, cardiovascular risk factors, and moderate to severely impaired renal function.

ELIGIBILITY:
Inclusion criteria :

* Type 2 Diabetes Mellitus with glycosylated hemoglobin (HbA1c) ≥7%.
* Estimated glomerular filtration rate (eGFR) ≥25 and ≤60 milliliter/minute (mL/min)/1.73 square meter (m^2).
* Age 18 years or older with at least one major cardiovascular risk factor or age 55 years or older with at least two minor cardiovascular risk factors.
* Signed written informed consent.

Exclusion criteria:

* Antihyperglycemic treatment has not been stable within 12 weeks prior to screening.
* Planned coronary procedure or surgery after randomization.
* Lower extremity complications (such as skin ulcer, infection, osteomyelitis, and gangrene) identified during screening and requiring treatment at randomization.
* Planning to start a sodium-glucose linked transporter-2 (SGLT2) inhibitor during the study.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10584 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (754):
- United States (119):
  - Investigational Site Number 8400017, Birmingham, Alabama
  - Investigational Site Number 8400096, Sheffield, Alabama
  - Investigational Site Number 8400004, Mesa, Arizona
  - Investigational Site Number 8400059, Mesa, Arizona
  - Investigational Site Number 8400021, Peoria, Arizona
  - Investigational Site Number 8400014, Surprise, Arizona
  - Investigational Site Number 8400071, Little Rock, Arkansas
  - Investigational Site Number 8400039, Beverly Hills, California
  - Investigational Site Number 8400042, Concord, California
  - Investigational Site Number 8400089, Fresno, California
  - Investigational Site Number 8400006, Huntington Park, California
  - Investigational Site Number 8400036, Long Beach, California
  - Investigational Site Number 8400073, Los Angeles, California
  - Investigational Site Number 8400084, Los Angeles, California
  - Investigational Site Number 8400035, Los Gatos, California
  - Investigational Site Number 8400043, Northridge, California
  - Investigational Site Number 8400025, Sacramento, California
  - Investigational Site Number 8400018, San Dimas, California
  - Investigational Site Number 8400070, Temecula, California
  - Investigational Site Number 8400013, Waterbury, Connecticut
  - Investigational Site Number 8400095, Bradenton, Florida
  - Investigational Site Number 8400090, Clearwater, Florida
  - Investigational Site Number 8400121, Clearwater, Florida
  - Investigational Site Number 8400049, Cooper City, Florida
  - Investigational Site Number 8400092, Hialeah, Florida
  - Investigational Site Number 8400026, Hollywood, Florida
  - Investigational Site Number 8400134, Jacksonville, Florida
  - Investigational Site Number 8400055, Jacksonville, Florida
  - Investigational Site Number 8400056, Jacksonville, Florida
  - Investigational Site Number 8400031, Jacksonville, Florida
  - Investigational Site Number 8400037, Maitland, Florida
  - Investigational Site Number 8400078, Miami, Florida
  - Investigational Site Number 8400117, Miami, Florida
  - Investigational Site Number 8400119, Miami, Florida
  - Investigational Site Number 8400118, Miami, Florida
  - Investigational Site Number 8400105, Miami, Florida
  - Investigational Site Number 8400120, Miami, Florida
  - Investigational Site Number 8400088, North Miami Beach, Florida
  - Investigational Site Number 8400106, Opa-locka, Florida
  - Investigational Site Number 8400063, Ormond Beach, Florida
  - Investigational Site Number 8400087, Palm Harbor, Florida
  - Investigational Site Number 8400108, Spring Hill, Florida
  - Investigational Site Number 8400058, St. Petersburg, Florida
  - Investigational Site Number 8400051, Tampa, Florida
  - Investigational Site Number 8400123, Atlanta, Georgia
  - Investigational Site Number 8400076, Roswell, Georgia
  - Investigational Site Number 8400033, Honolulu, Hawaii
  - Investigational Site Number 8400085, Arlington Heights, Illinois
  - Investigational Site Number 8400104, Chicago, Illinois
  - Investigational Site Number 8400027, Chicago, Illinois
  - Investigational Site Number 8400124, Chicago, Illinois
  - Investigational Site Number 8400001, Chicago, Illinois
  - Investigational Site Number 8400052, Crystal Lake, Illinois
  - Investigational Site Number 8400028, Springfield, Illinois
  - Investigational Site Number 8400125, Michigan City, Indiana
  - Investigational Site Number 8400098, Valparaiso, Indiana
  - Investigational Site Number 8400003, Des Moines, Iowa
  - Investigational Site Number 8400081, Topeka, Kansas
  - Investigational Site Number 8400041, Louisville, Kentucky
  - Investigational Site Number 8400080, Bangor, Maine
  - Investigational Site Number 8400002, Flint, Michigan
  - Investigational Site Number 8400069, Flint, Michigan
  - Investigational Site Number 8400016, Troy, Michigan
  - Investigational Site Number 8400023, Saint Cloud, Minnesota
  - Investigational Site Number 8400066, Kansas City, Missouri
  - Investigational Site Number 8400024, St Louis, Missouri
  - Investigational Site Number 8400130, Washington, Missouri
  - Investigational Site Number 8400045, Omaha, Nebraska
  - Investigational Site Number 8400009, Las Vegas, Nevada
  - Investigational Site Number 8400101, Albany, New York
  - Investigational Site Number 8400061, Laurelton, New York
  - Investigational Site Number 8400046, New York, New York
  - Investigational Site Number 8400112, Rosedale, New York
  - Investigational Site Number 8400062, Smithtown, New York
  - Investigational Site Number 8400079, Greenville, North Carolina
  - Investigational Site Number 8400020, Morehead City, North Carolina
  - Investigational Site Number 8400048, Morehead City, North Carolina
  - Investigational Site Number 8400010, Morganton, North Carolina
  - Investigational Site Number 8400072, Fargo, North Dakota
  - Investigational Site Number 8400038, Cincinnati, Ohio
  - Investigational Site Number 8400007, Cincinnati, Ohio
  - Investigational Site Number 8400015, Columbus, Ohio
  - Investigational Site Number 8400113, Lorain, Ohio
  - Investigational Site Number 8400011, Mentor, Ohio
  - Investigational Site Number 8400109, Bend, Oregon
  - Investigational Site Number 8400047, Beaver, Pennsylvania
  - Investigational Site Number 8400019, Greensburg, Pennsylvania
  - Investigational Site Number 8400097, Indiana, Pennsylvania
  - Investigational Site Number 8400032, Levittown, Pennsylvania
  - Investigational Site Number 8400053, Philadelphia, Pennsylvania
  - Investigational Site Number 8400012, Pittsburgh, Pennsylvania
  - Investigational Site Number 8400064, Anderson, South Carolina
  - Investigational Site Number 8400030, Greer, South Carolina
  - Investigational Site Number 8400029, Myrtle Beach, South Carolina
  - Investigational Site Number 8400040, Memphis, Tennessee
  - Investigational Site Number 8400114, Arlington, Texas
  - Investigational Site Number 8400067, Corpus Christi, Texas
  - Investigational Site Number 8400082, Dallas, Texas
  - Investigational Site Number 8400022, El Paso, Texas
  - Investigational Site Number 8400099, Houston, Texas
  - Investigational Site Number 8400103, Houston, Texas
  - Investigational Site Number 8400086, Katy, Texas
  - Investigational Site Number 8400100, Mesquite, Texas
  - Investigational Site Number 8400094, Plano, Texas
  - Investigational Site Number 8400116, San Antonio, Texas
  - Investigational Site Number 8400091, Waco, Texas
  - Investigational Site Number 8400065, Bountiful, Utah
  - Investigational Site Number 8400131, Ogden, Utah
  - Investigational Site Number 8400093, Bennington, Vermont
  - Investigational Site Number 8400060, South Burlington, Vermont
  - Investigational Site Number 8400133, Danville, Virginia
  - Investigational Site Number 8400054, Fairfax, Virginia
  - Investigational Site Number 8400132, Falls Church, Virginia
  - Investigational Site Number 8400034, Manassas, Virginia
  - Investigational Site Number 8400050, Norfolk, Virginia
  - Investigational Site Number 8400044, Richmond, Virginia
  - Investigational Site Number 8400111, Richmond, Virginia
  - Investigational Site Number 8400083, Federal Way, Washington
  - Investigational Site Number 8400068, Spokane, Washington
- Argentina (29):
  - Investigational Site Number 0320016, Buenos Aires
  - Investigational Site Number 0320029, Buenos Aires
  - Investigational Site Number 0320017, Caba
  - Investigational Site Number 0320002, Caba
  - Investigational Site Number 0320004, Caba
  - Investigational Site Number 0320018, Caba
  - Investigational Site Number 0320025, Caba
  - Investigational Site Number 0320019, Caba
  - Investigational Site Number 0320027, Capital Federal
  - Investigational Site Number 0320015, Capital Federal
  - Investigational Site Number 0320014, Ciudad Autonoma de Bs.As
  - Investigational Site Number 0320023, Ciudad Autonoma de Buenos Aire
  - Investigational Site Number 0320009, Ciudadela
  - Investigational Site Number 0320008, Coronel Suárez
  - Investigational Site Number 0320011, Corrientes
  - Investigational Site Number 0320001, Córdoba
  - Investigational Site Number 0320028, La Plata
  - Investigational Site Number 0320006, La Plata
  - Investigational Site Number 0320024, Mar del Plata
  - Investigational Site Number 0320003, Mar del Plata
  - Investigational Site Number 0320020, Merlo
  - Investigational Site Number 0320007, Ramos Mejía
  - Investigational Site Number 0320030, Rosario
  - Investigational Site Number 0320026, Rosario
  - Investigational Site Number 0320012, Salta
  - Investigational Site Number 0320021, San Miguel de Tucumán
  - Investigational Site Number 0320013, Santa Fe
  - Investigational Site Number 0320022, Temperley
  - Investigational Site Number 0320005, Villa María
- Australia (18):
  - Investigational Site Number 0360014, Adelaide
  - Investigational Site Number 0360004, Box Hill
  - Investigational Site Number 0360015, Elizabeth Vale
  - Investigational Site Number 0360005, Fitzroy
  - Investigational Site Number 0360018, Fremantle
  - Investigational Site Number 0360007, Fullarton
  - Investigational Site Number 0360002, Gosford
  - Investigational Site Number 0360016, Heidelberg
  - Investigational Site Number 0360010, Herston
  - Investigational Site Number 0360009, Liverpool
  - Investigational Site Number 0360017, Melbourne
  - Investigational Site Number 0360001, Merewether
  - Investigational Site Number 0360012, Oaklands Park
  - Investigational Site Number 0360011, Parkville
  - Investigational Site Number 0360008, Redcliffe
  - Investigational Site Number 0360013, Sherwood
  - Investigational Site Number 0360019, St Leonards
  - Investigational Site Number 0360006, Wollongong
- Belgium (5):
  - Investigational Site Number 0560004, Bonheiden
  - Investigational Site Number 0560005, Ghent
  - Investigational Site Number 0560003, Kortrijk
  - Investigational Site Number 0560002, La Louvière
  - Investigational Site Number 0560001, Leuven
- Brazil (26):
  - Investigational Site Number 0760017, Blumenau
  - Investigational Site Number 0760015, Brasília
  - Investigational Site Number 0760026, Brasília
  - Investigational Site Number 0760008, Campinas
  - Investigational Site Number 0760005, Campinas
  - Investigational Site Number 0760018, Canoas
  - Investigational Site Number 0760019, Curitiba
  - Investigational Site Number 0760011, Curitiba
  - Investigational Site Number 0760007, Curitiba
  - Investigational Site Number 0760010, Fortaleza
  - Investigational Site Number 0760002, Fortaleza
  - Investigational Site Number 0760004, Fortaleza
  - Investigational Site Number 0760014, Passo Fundo
  - Investigational Site Number 0760025, Porto Alegre
  - Investigational Site Number 0760016, Porto Alegre
  - Investigational Site Number 0760024, Recife
  - Investigational Site Number 0760023, Rio de Janeiro
  - Investigational Site Number 0760001, São José do Rio Preto
  - Investigational Site Number 0760012, São José dos Campos
  - Investigational Site Number 0760003, São Paulo
  - Investigational Site Number 0760020, São Paulo
  - Investigational Site Number 0760013, São Paulo
  - Investigational Site Number 0760022, São Paulo
  - Investigational Site Number 0760006, São Paulo
  - Investigational Site Number 0760009, São Paulo
  - Investigational Site Number 0760021, Vitória
- Bulgaria (15):
  - Investigational Site Number 1000015, Blagoevgrad
  - Investigational Site Number 1000008, Dobrich
  - Investigational Site Number 1000013, Gabrovo
  - Investigational Site Number 1000003, Plovdiv
  - Investigational Site Number 1000016, Rousse
  - Investigational Site Number 1000014, Silistra
  - Investigational Site Number 1000007, Smolyan
  - Investigational Site Number 1000011, Sofia
  - Investigational Site Number 1000004, Sofia
  - Investigational Site Number 1000006, Sofia
  - Investigational Site Number 1000012, Sofia
  - Investigational Site Number 1000005, Sofia
  - Investigational Site Number 1000017, Sofia
  - Investigational Site Number 1000001, Stara Zagora
  - Investigational Site Number 1000018, Stara Zagora
- Canada (30):
  - Investigational Site Number 1240002, Brampton
  - Investigational Site Number 1240013, Burlington
  - Investigational Site Number 1240021, Calgary
  - Investigational Site Number 1240005, Calgary
  - Investigational Site Number 1240029, Concord
  - Investigational Site Number 1240004, Edmonton
  - Investigational Site Number 1240010, Edmonton
  - Investigational Site Number 1240008, Greater Sudbury
  - Investigational Site Number 1240027, Halifax
  - Investigational Site Number 1240023, Hamilton
  - Investigational Site Number 1240011, London
  - Investigational Site Number 1240019, Montreal
  - Investigational Site Number 1240017, Montreal
  - Investigational Site Number 1240018, Montreal
  - Investigational Site Number 1240007, Newmarket
  - Investigational Site Number 1240026, Oshawa
  - Investigational Site Number 1240016, Oshawa
  - Investigational Site Number 1240006, Ottawa
  - Investigational Site Number 1240022, Québec
  - Investigational Site Number 1240025, Québec
  - Investigational Site Number 1240014, Québec
  - Investigational Site Number 1240003, Québec
  - Investigational Site Number 1240034, Saint-Charles-Borromée
  - Investigational Site Number 1240032, Saint-Marc-des-Carrieres
  - Investigational Site Number 1240033, St. John's
  - Investigational Site Number 1240031, Surrey
  - Investigational Site Number 1240028, Toronto
  - Investigational Site Number 1240015, Trois-Rivières
  - Investigational Site Number 1240001, Vancouver
  - Investigational Site Number 1240030, Victoria
- Chile (25):
  - Investigational Site Number 1520015, Concepción
  - Investigational Site Number 1520003, Osorno
  - Investigational Site Number 1520012, Punta Arenas
  - Investigational Site Number 1520013, Santiago
  - Investigational Site Number 1520018, Santiago
  - Investigational Site Number 1520001, Santiago
  - Investigational Site Number 1520004, Santiago
  - Investigational Site Number 1520006, Santiago
  - Investigational Site Number 1520014, Santiago
  - Investigational Site Number 1520016, Santiago
  - Investigational Site Number 1520017, Santiago
  - Investigational Site Number 1520020, Santiago
  - Investigational Site Number 1520009, Santiago
  - Investigational Site Number 1520011, Santiago
  - Investigational Site Number 1520026, Santiago
  - Investigational Site Number 1520010, Santiago
  - Investigational Site Number 1520007, Santiago
  - Investigational Site Number 1520021, Santiago
  - Investigational Site Number 1520022, Santiago
  - Investigational Site Number 1520002, Santiago
  - Investigational Site Number 1520024, Talca
  - Investigational Site Number 1520019, Temuco
  - Investigational Site Number 1520025, Temuco
  - Investigational Site Number 1520005, Temuco
  - Investigational Site Number 1520008, Viña del Mar
- China (33):
  - Investigational Site Number 1560019, Beijing
  - Investigational Site Number 1560001, Beijing
  - Investigational Site Number 1560002, Beijing
  - Investigational Site Number 1560003, Beijing
  - Investigational Site Number 1560032, Beijing
  - Investigational Site Number 1560012, Changchun
  - Investigational Site Number 1560023, Changchun
  - Investigational Site Number 1560034, Changchun
  - Investigational Site Number 1560022, Changsha
  - Investigational Site Number 1560021, Chengdu
  - Investigational Site Number 1560018, Dalian
  - Investigational Site Number 1560010, Dalian
  - Investigational Site Number 1560007, Guangzhou
  - Investigational Site Number 1560016, Haikou
  - Investigational Site Number 1560033, Hengyang
  - Investigational Site Number 1560038, Hohhot
  - Investigational Site Number 1560005, Huai'an
  - Investigational Site Number 1560009, Jinan
  - Investigational Site Number 1560037, Jining
  - Investigational Site Number 1560031, Nanchang
  - Investigational Site Number 1560004, Nanjing
  - Investigational Site Number 1560006, Shanghai
  - Investigational Site Number 1560036, Shenyang
  - Investigational Site Number 1560020, Siping
  - Investigational Site Number 1560025, Suzhou
  - Investigational Site Number 1560014, Suzhou
  - Investigational Site Number 1560026, Taizhou
  - Investigational Site Number 1560028, Tianjin
  - Investigational Site Number 1560029, Tianjin
  - Investigational Site Number 1560024, Wuhan
  - Investigational Site Number 1560027, Xi'an
  - Investigational Site Number 1560035, Xinxiang
  - Investigational Site Number 1560008, Zhenjiang
- Czechia (18):
  - Investigational Site Number 2030012, Brno
  - Investigational Site Number 2030002, Brno
  - Investigational Site Number 2030021, Broumov
  - Investigational Site Number 2030017, Humpolec
  - Investigational Site Number 2030014, Liberec
  - Investigational Site Number 2030007, Mariánské Lázně
  - Investigational Site Number 2030015, Městec Králové
  - Investigational Site Number 2030009, Pilsen
  - Investigational Site Number 2030016, Prague
  - Investigational Site Number 2030019, Prague
  - Investigational Site Number 2030006, Prague
  - Investigational Site Number 2030005, Prague
  - Investigational Site Number 2030011, Prague
  - Investigational Site Number 2030018, Prague
  - Investigational Site Number 2030010, Řevnice
  - Investigational Site Number 2030020, Slaný
  - Investigational Site Number 2030001, Trutnov
  - Investigational Site Number 2030008, Vsetín
- Denmark (8):
  - Investigational Site Number 2080003, Aarhus N
  - Investigational Site Number 2080005, Aarhus N
  - Investigational Site Number 2080009, Gentofte Municipality
  - Investigational Site Number 2080004, Herlev
  - Investigational Site Number 2080008, Hvidovre
  - Investigational Site Number 2080002, København NV
  - Investigational Site Number 2080007, Slagelse
  - Investigational Site Number 2080006, Svendborg
- Estonia (3):
  - Investigational Site Number 2330003, Tallinn
  - Investigational Site Number 2330001, Tallinn
  - Investigational Site Number 2330002, Tartu
- France (7):
  - Investigational Site Number 2500003, Corbeil-Essonnes
  - Investigational Site Number 2500002, La Rochelle
  - Investigational Site Number 2500005, Paris
  - Investigational Site Number 2500006, Paris
  - Investigational Site Number 2500001, Paris
  - Investigational Site Number 2500004, Toulouse
  - Investigational Site Number 2500007, Vénissieux
- Georgia (7):
  - Investigational Site Number 2680004, Batumi
  - Investigational Site Number 2680001, Kutaisi
  - Investigational Site Number 2680007, Tbilisi
  - Investigational Site Number 2680005, Tbilisi
  - Investigational Site Number 2680003, Tbilisi
  - Investigational Site Number 2680006, Tbilisi
  - Investigational Site Number 2680002, Tbilisi
- Germany (8):
  - Investigational Site Number 2760008, Berlin
  - Investigational Site Number 2760005, Essen
  - Investigational Site Number 2760001, Freiburg im Breisgau
  - Investigational Site Number 2760007, Hamburg
  - Investigational Site Number 2760002, Kassel
  - Investigational Site Number 2760006, Leipzig
  - Investigational Site Number 2760003, Münster
  - Investigational Site Number 2760009, Oldenburg in Holstein
- Greece (5):
  - Investigational Site Number 3000001, Athens
  - Investigational Site Number 3000002, Ioannina
  - Investigational Site Number 3000004, Larissa
  - Investigational Site Number 3000003, Piraeus
  - Investigational Site Number 3000005, Thessaloniki
- Guatemala (9):
  - Investigational Site Number 3200007, Guatemala City
  - Investigational Site Number 3200013, Guatemala City
  - Investigational Site Number 3200001, Guatemala City
  - Investigational Site Number 3200002, Guatemala City
  - Investigational Site Number 3200009, Guatemala City
  - Investigational Site Number 3200010, Guatemala City
  - Investigational Site Number 3200006, Quetzaltenango
  - Investigational Site Number 3200014, Quetzaltenango
  - Investigational Site Number 3200004, Quetzaltenango
- Hungary (16):
  - Investigational Site Number 3480006, Békéscsaba
  - Investigational Site Number 3480017, Budapest
  - Investigational Site Number 3480004, Budapest
  - Investigational Site Number 3480011, Budapest
  - Investigational Site Number 3480001, Budapest
  - Investigational Site Number 3480010, Budapest
  - Investigational Site Number 3480012, Budapest
  - Investigational Site Number 3480016, Budapest
  - Investigational Site Number 3480018, Budapest
  - Investigational Site Number 3480002, Debrecen
  - Investigational Site Number 3480008, Debrecen
  - Investigational Site Number 3480013, Kaposvár
  - Investigational Site Number 3480014, Nyíregyháza
  - Investigational Site Number 3480015, Nyíregyháza
  - Investigational Site Number 3480003, Székesfehérvár
  - Investigational Site Number 3480007, Zalaegerszeg
- India (34):
  - Investigational Site Number 3560025, Ahmedabad
  - Investigational Site Number 3560040, Aurangabad
  - Investigational Site Number 3560010, Bangalore
  - Investigational Site Number 3560026, Bangalore
  - Investigational Site Number 3560005, Belagavi
  - Investigational Site Number 3560008, Bengaluru
  - Investigational Site Number 3560022, Chandigarh
  - Investigational Site Number 3560003, Gūrgaon
  - Investigational Site Number 3560004, Gūrgaon
  - Investigational Site Number 3560018, Hyderabad
  - Investigational Site Number 3560001, Hyderabad
  - Investigational Site Number 3560007, Hyderabad
  - Investigational Site Number 3560002, Jaipur
  - Investigational Site Number 3560024, Kochi
  - Investigational Site Number 3560016, Kolkata
  - Investigational Site Number 3560030, Kozhikode
  - Investigational Site Number 3560006, Ludhiana
  - Investigational Site Number 3560027, Mangalore
  - Investigational Site Number 3560028, Mangalore
  - Investigational Site Number 3560017, Mumbai
  - Investigational Site Number 3560037, Mysore
  - Investigational Site Number 3560013, Nagpur
  - Investigational Site Number 3560014, Nagpur
  - Investigational Site Number 3560021, Nashik
  - Investigational Site Number 3560041, New Delhi
  - Investigational Site Number 3560034, New Delhi
  - Investigational Site Number 3560019, Pune
  - Investigational Site Number 3560035, Pune
  - Investigational Site Number 3560042, Pune
  - Investigational Site Number 3560038, Pune
  - Investigational Site Number 3560012, Pune
  - Investigational Site Number 3560043, Varanasi
  - Investigational Site Number 3560020, Vellore
  - Investigational Site Number 3560015, Wardha
- Israel (8):
  - Investigational Site Number 3760008, Beersheba
  - Investigational Site Number 3760005, Haifa
  - Investigational Site Number 3760007, Haifa
  - Investigational Site Number 3760001, Jerusalem
  - Investigational Site Number 3760002, Jerusalem
  - Investigational Site Number 3760004, Nahariya
  - Investigational Site Number 3760003, Tel Aviv
  - Investigational Site Number 3760006, Tel Litwinsky
- Italy (10):
  - Investigational Site Number 3800006, Catanzaro
  - Investigational Site Number 3800010, Catanzaro
  - Investigational Site Number 3800009, Chieri
  - Investigational Site Number 3800007, Livorno
  - Investigational Site Number 3800002, Milan
  - Investigational Site Number 3800008, Milan
  - Investigational Site Number 3800005, Orbassano
  - Investigational Site Number 3800011, Ravenna
  - Investigational Site Number 3800004, Roma
  - Investigational Site Number 3800001, Verona
- Latvia (7):
  - Investigational Site Number 4280004, Daugavpils
  - Investigational Site Number 4280002, Liepāja
  - Investigational Site Number 4280007, Ogre
  - Investigational Site Number 4280006, Riga
  - Investigational Site Number 4280001, Riga
  - Investigational Site Number 4280005, Riga
  - Investigational Site Number 4280003, Sigulda
- Lithuania (9):
  - Investigational Site Number 4400006, Kaunas
  - Investigational Site Number 4400003, Kaunas
  - Investigational Site Number 4400009, Kaunas
  - Investigational Site Number 4400008, Kėdainiai
  - Investigational Site Number 4400004, Klaipėda
  - Investigational Site Number 4400002, Klaipėda
  - Investigational Site Number 4400007, Ukmerge
  - Investigational Site Number 4400005, Utena
  - Investigational Site Number 4400001, Vilnius
- Mexico (27):
  - Investigational Site Number 4840009, Actopan
  - Investigational Site Number 4840013, Aguascalientes
  - Investigational Site Number 4840019, Aguascalientes
  - Investigational Site Number 4840005, Celaya
  - Investigational Site Number 4840002, Cuernavaca
  - Investigational Site Number 4840025, Distrito Federal
  - Investigational Site Number 4840007, Durango
  - Investigational Site Number 4840023, Durango
  - Investigational Site Number 4840033, Guadalajara
  - Investigational Site Number 4840024, Guadalajara
  - Investigational Site Number 4840003, Guadalajara
  - Investigational Site Number 4840011, Guadalajara
  - Investigational Site Number 4840027, Guadalajara
  - Investigational Site Number 4840004, Guadalajara
  - Investigational Site Number 4840010, Guadalajara
  - Investigational Site Number 4840030, Guadalajara
  - Investigational Site Number 4840018, Mexico City
  - Investigational Site Number 4840028, Mérida
  - Investigational Site Number 4840034, Mérida
  - Investigational Site Number 4840021, Monterrey
  - Investigational Site Number 4840020, Monterrey
  - Investigational Site Number 4840001, Monterrey
  - Investigational Site Number 4840014, Querétaro
  - Investigational Site Number 4840015, Toluca
  - Investigational Site Number 4840008, Veracruz
  - Investigational Site Number 4840016, Xalapa
  - Investigational Site Number 4840026, Zapopan
- Netherlands (5):
  - Investigational Site Number 5280004, Almelo
  - Investigational Site Number 5280001, Groningen
  - Investigational Site Number 5280003, Hoogeveen
  - Investigational Site Number 5280005, Meppel
  - Investigational Site Number 5280002, Rotterdam
- New Zealand (15):
  - Investigational Site Number 5540014, Auckland
  - Investigational Site Number 5540006, Birkenhead
  - Investigational Site Number 5540009, Birkenhead
  - Investigational Site Number 5540002, Christchurch
  - Investigational Site Number 5540003, Christchurch
  - Investigational Site Number 5540012, Christchurch
  - Investigational Site Number 5540007, Dunedin
  - Investigational Site Number 5540016, Hamilton
  - Investigational Site Number 5540013, New Plymouth
  - Investigational Site Number 5540015, Palmerston North
  - Investigational Site Number 5540005, Rotorua
  - Investigational Site Number 5540010, Takapuna
  - Investigational Site Number 5540008, Tauranga
  - Investigational Site Number 5540011, Tauranga
  - Investigational Site Number 5540004, Wellington
- North Macedonia (4):
  - Investigational Site Number 8070003, Skopje
  - Investigational Site Number 8070005, Struga
  - Investigational Site Number 8070001, Tetovo
  - Investigational Site Number 8070004, Tetovo
- Norway (5):
  - Investigational Site Number 5780005, Hamar
  - Investigational Site Number 5780001, Hønefoss
  - Investigational Site Number 5780003, Oslo
  - Investigational Site Number 5780002, Oslo
  - Investigational Site Number 5780004, Skedsmokorset
- Peru (20):
  - Investigational Site Number 6040004, Arequipa
  - Investigational Site Number 6040006, Callao
  - Investigational Site Number 6040009, Callao
  - Investigational Site Number 6040024, Chancay
  - Investigational Site Number 6040005, Chiclayo
  - Investigational Site Number 6040010, Cuzco
  - Investigational Site Number 6040001, Lima
  - Investigational Site Number 6040025, Lima
  - Investigational Site Number 6040016, Lima
  - Investigational Site Number 6040020, Lima
  - Investigational Site Number 6040013, Lima
  - Investigational Site Number 6040023, Lima
  - Investigational Site Number 6040007, Lima
  - Investigational Site Number 6040019, Lima
  - Investigational Site Number 6040022, Lima
  - Investigational Site Number 6040012, Lima
  - Investigational Site Number 6040017, Lima
  - Investigational Site Number 6040014, Lima Lima
  - Investigational Site Number 6040011, Piura
  - Investigational Site Number 6040002, Trujillo
- Poland (32):
  - Investigational Site Number 6160027, Bialystok
  - Investigational Site Number 6160011, Bialystok
  - Investigational Site Number 6160029, Bydgoszcz
  - Investigational Site Number 6160030, Bydgoszcz
  - Investigational Site Number 6160006, Bydgoszcz
  - Investigational Site Number 6160018, Bytom
  - Investigational Site Number 6160002, Czeladź
  - Investigational Site Number 6160003, Gdynia
  - Investigational Site Number 6160005, Gdynia
  - Investigational Site Number 6160008, Grodzisk Mazowiecki
  - Investigational Site Number 6160031, Grodzisk Mazowiecki
  - Investigational Site Number 6160023, Katowice
  - Investigational Site Number 6160026, Katowice
  - Investigational Site Number 6160022, Kielce
  - Investigational Site Number 6160019, Krakow
  - Investigational Site Number 6160024, Krakow
  - Investigational Site Number 6160010, Krakow
  - Investigational Site Number 6160016, Lodz
  - Investigational Site Number 6160013, Lodz
  - Investigational Site Number 6160015, Lodz
  - Investigational Site Number 6160007, Lublin
  - Investigational Site Number 6160033, Poznan
  - Investigational Site Number 6160021, Puławy
  - Investigational Site Number 6160028, Staszów
  - Investigational Site Number 6160020, Torun
  - Investigational Site Number 6160014, Warsaw
  - Investigational Site Number 6160025, Warsaw
  - Investigational Site Number 6160001, Warsaw
  - Investigational Site Number 6160004, Warsaw
  - Investigational Site Number 6160012, Wroclaw
  - Investigational Site Number 6160017, Zabrze
  - Investigational Site Number 6160032, Zamość
- Portugal (8):
  - Investigational Site Number 6200004, Almada
  - Investigational Site Number 6200005, Caldas da Rainha
  - Investigational Site Number 6200009, Carnaxide
  - Investigational Site Number 6200002, Coimbra
  - Investigational Site Number 6200008, Leiria
  - Investigational Site Number 6200001, Lisbon
  - Investigational Site Number 6200007, Loures
  - Investigational Site Number 6200003, Porto
- Investigational Site Number 8400122, San Juan, Puerto Rico
- Romania (14):
  - Investigational Site Number 6420008, Bacau
  - Investigational Site Number 6420005, Baia Mare, Maramures
  - Investigational Site Number 6420009, Brasov
  - Investigational Site Number 6420013, Bucharest
  - Investigational Site Number 6420014, Bucharest
  - Investigational Site Number 6420012, Bucharest
  - Investigational Site Number 6420011, Bucharest
  - Investigational Site Number 6420002, Craiova
  - Investigational Site Number 6420003, Oradea
  - Investigational Site Number 6420004, Oradea
  - Investigational Site Number 6420010, Ploieşti
  - Investigational Site Number 6420001, Targoviste, Dambovita
  - Investigational Site Number 6420006, Targu Mures, Mures
  - Investigational Site Number 6420007, Targu Mures, Mures
- Russia (45):
  - Investigational Site Number 6430028, Kaliningrad
  - Investigational Site Number 6430018, Kazan'
  - Investigational Site Number 6430001, Kemerovo
  - Investigational Site Number 6430035, Kemerovo
  - Investigational Site Number 6430025, Krasnodar
  - Investigational Site Number 6430040, Krasnodar
  - Investigational Site Number 6430010, Krasnodar
  - Investigational Site Number 6430015, Moscow
  - Investigational Site Number 6430016, Moscow
  - Investigational Site Number 6430046, Moscow
  - Investigational Site Number 6430003, Moscow
  - Investigational Site Number 6430036, Moscow
  - Investigational Site Number 6430005, Moscow
  - Investigational Site Number 6430039, Moscow
  - Investigational Site Number 6430021, Moscow
  - Investigational Site Number 6430002, Moscow
  - Investigational Site Number 6430020, Moscow
  - Investigational Site Number 6430024, Moscow
  - Investigational Site Number 6430033, Nizhny Novgorod
  - Investigational Site Number 6430037, Novosibirsk
  - Investigational Site Number 6430034, Novosibirsk
  - Investigational Site Number 6430007, Perm
  - Investigational Site Number 6430019, Rostov-on-Don
  - Investigational Site Number 6430012, Saint Petersburg
  - Investigational Site Number 6430041, Saint Petersburg
  - Investigational Site Number 6430006, Saint Petersburg
  - Investigational Site Number 6430008, Saint Petersburg
  - Investigational Site Number 6430030, Saint Petersburg
  - Investigational Site Number 6430044, Saint Petersburg
  - Investigational Site Number 6430045, Saint Petersburg
  - Investigational Site Number 6430014, Saint Petersburg
  - Investigational Site Number 6430017, Saint Petersburg
  - Investigational Site Number 6430043, Saint Petersburg
  - Investigational Site Number 6430004, Saint Petersburg
  - Investigational Site Number 6430009, Saratov
  - Investigational Site Number 6430013, Saratov
  - Investigational Site Number 6430042, Saratov
  - Investigational Site Number 6430026, Sochi
  - Investigational Site Number 6430027, Sochi
  - Investigational Site Number 6430011, Tomsk
  - Investigational Site Number 6430038, Tomsk
  - Investigational Site Number 6430032, Tyumen
  - Investigational Site Number 6430023, Vladimir
  - Investigational Site Number 6430022, Vladimir
  - Investigational Site Number 6430031, Yaroslavl
- Serbia (7):
  - Investigational Site Number 6880002, Belgrade
  - Investigational Site Number 6880003, Belgrade
  - Investigational Site Number 6880004, Belgrade
  - Investigational Site Number 6880005, Kragujevac
  - Investigational Site Number 6880001, Niš
  - Investigational Site Number 6880006, Niš
  - Investigational Site Number 6880007, Niš
- Slovakia (12):
  - Investigational Site Number 7030006, Bardejov
  - Investigational Site Number 7030012, Bratislava
  - Investigational Site Number 7030011, Košice
  - Investigational Site Number 7030008, Lučenec
  - Investigational Site Number 7030009, Lučenec
  - Investigational Site Number 7030010, Lučenec
  - Investigational Site Number 7030001, Ľubochňa
  - Investigational Site Number 7030004, Moldava nad Bodvou
  - Investigational Site Number 7030013, Prešov
  - Investigational Site Number 7030003, Rožňava
  - Investigational Site Number 7030002, Sabinov
  - Investigational Site Number 7030007, Svidník
- South Africa (13):
  - Investigational Site Number 7100005, Brits
  - Investigational Site Number 7100009, Cape Town
  - Investigational Site Number 7100006, Cape Town
  - Investigational Site Number 7100002, eMkhomazi
  - Investigational Site Number 7100001, Parow
  - Investigational Site Number 7100012, Pinelands
  - Investigational Site Number 7100011, Pretoria
  - Investigational Site Number 7100014, Pretoria
  - Investigational Site Number 7100008, Pretoria
  - Investigational Site Number 7100010, Rivonia
  - Investigational Site Number 7100007, Soweto
  - Investigational Site Number 7100013, Vosloorus
  - Investigational Site Number 7100003, Western Cape
- South Korea (10):
  - Investigational Site Number 4100011, Bucheon-si
  - Investigational Site Number 4100005, Busan
  - Investigational Site Number 4100007, Gwangju
  - Investigational Site Number 4100001, Incheon
  - Investigational Site Number 4100002, Seongnam-si
  - Investigational Site Number 4100003, Seoul
  - Investigational Site Number 4100006, Seoul
  - Investigational Site Number 4100008, Seoul
  - Investigational Site Number 4100004, Seoul
  - Investigational Site Number 4100010, Uijeongbu-si
- Spain (22):
  - Investigational Site Number 7240015, A Coruña
  - Investigational Site Number 7240003, Almería
  - Investigational Site Number 7240014, Barcelona
  - Investigational Site Number 7240011, Barcelona
  - Investigational Site Number 7240009, Córdoba
  - Investigational Site Number 7240024, El Puerto de Santa María
  - Investigational Site Number 7240016, Granada
  - Investigational Site Number 7240001, Madrid
  - Investigational Site Number 7240019, Madrid
  - Investigational Site Number 7240006, Madrid
  - Investigational Site Number 7240010, Madrid
  - Investigational Site Number 7240020, Madrid
  - Investigational Site Number 7240025, Sabadell
  - Investigational Site Number 7240023, Sanlúcar de Barrameda
  - Investigational Site Number 7240013, Santa Cruz de Tenerife
  - Investigational Site Number 7240007, Santiago de Compostela
  - Investigational Site Number 7240026, Seville
  - Investigational Site Number 7240012, Seville
  - Investigational Site Number 7240004, Valencia
  - Investigational Site Number 7240002, Vigo
  - Investigational Site Number 7240022, Villamartín
  - Investigational Site Number 7240008, Zaragoza
- Sweden (8):
  - Investigational Site Number 7520007, Falun
  - Investigational Site Number 7520005, Lund
  - Investigational Site Number 7520004, Mölndal
  - Investigational Site Number 7520003, Rättvik
  - Investigational Site Number 7520008, Stockholm
  - Investigational Site Number 7520002, Stockholm
  - Investigational Site Number 7520006, Stockholm
  - Investigational Site Number 7520001, Uppsala
- Switzerland (2):
  - Investigational Site Number 7560001, Olten
  - Investigational Site Number 7560002, Zollikerberg
- Taiwan (8):
  - Investigational Site Number 1580005, Hsinchu
  - Investigational Site Number 1580008, Kaohsiung City
  - Investigational Site Number 1580004, Linkou District
  - Investigational Site Number 1580006, Taichung
  - Investigational Site Number 1580002, Tainan
  - Investigational Site Number 1580007, Tainan
  - Investigational Site Number 1580003, Taipei
  - Investigational Site Number 1580001, Taipei
- Turkey (Türkiye) (16):
  - Investigational Site Number 7920018, Antalya
  - Investigational Site Number 7920010, Aydin
  - Investigational Site Number 7920004, Çorum
  - Investigational Site Number 7920016, Gaziantep
  - Investigational Site Number 7920011, Istanbul
  - Investigational Site Number 7920009, Istanbul
  - Investigational Site Number 7920001, Istanbul
  - Investigational Site Number 7920007, Istanbul
  - Investigational Site Number 7920017, Istanbul
  - Investigational Site Number 7920003, Izmir
  - Investigational Site Number 7920013, Kayseri
  - Investigational Site Number 7920014, Kocaeli
  - Investigational Site Number 7920005, Kütahya
  - Investigational Site Number 7920015, Malatya
  - Investigational Site Number 7920008, Mersin
  - Investigational Site Number 7920002, Sivas
- Ukraine (22):
  - Investigational Site Number 8040020, Dnipro
  - Investigational Site Number 8040006, Dnipro
  - Investigational Site Number 8040009, Ivano-Frankivsk
  - Investigational Site Number 8040012, Ivano-Frankivsk
  - Investigational Site Number 8040021, Kharkiv
  - Investigational Site Number 8040011, Kharkiv
  - Investigational Site Number 8040008, Kharkiv
  - Investigational Site Number 8040002, Kiev
  - Investigational Site Number 8040024, Kiev
  - Investigational Site Number 8040003, Kyiv
  - Investigational Site Number 8040015, Kyiv
  - Investigational Site Number 8040019, Kyiv
  - Investigational Site Number 8040010, Kyiv
  - Investigational Site Number 8040026, Kyiv
  - Investigational Site Number 8040023, Lutsk
  - Investigational Site Number 8040025, Lutsk
  - Investigational Site Number 8040022, Lviv
  - Investigational Site Number 8040001, Ternopil
  - Investigational Site Number 8040016, Vinnitsya
  - Investigational Site Number 8040007, Vinnitsya
  - Investigational Site Number 8040004, Vinnytsia
  - Investigational Site Number 8040018, Zhytomyr
- United Kingdom (9):
  - Investigational Site Number 8260003, Belfast
  - Investigational Site Number 8260007, Chippenham
  - Investigational Site Number 8260009, Davyhulme, Manchester
  - Investigational Site Number 8260010, Glasgow
  - Investigational Site Number 8260004, Hayle
  - Investigational Site Number 8260011, Inverness
  - Investigational Site Number 8260002, Ipswich
  - Investigational Site Number 8260006, Maidstone
  - Investigational Site Number 8260001, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants.

REFERENCES:
- [Derived] Aggarwal R, Bhatt DL, Szarek M, Cannon CP, Leiter LA, Inzucchi SE, Lopes RD, McGuire DK, Lewis JB, Riddle MC, Davies MJ, Banks P, Carroll AK, Scirica BM, Ray KK, Kosiborod MN, Cherney DZI, Udell JA, Verma S, Mason RP, Pitt B, Steg PG. Effect of sotagliflozin on major adverse cardiovascular events: a prespecified secondary analysis of the SCORED randomised trial. Lancet Diabetes Endocrinol. 2025 Apr;13(4):321-332. doi: 10.1016/S2213-8587(24)00362-0. Epub 2025 Feb 14. PMID 39961315
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Sridhar VS, Bhatt DL, Odutayo A, Szarek M, Davies MJ, Banks P, Pitt B, Steg PG, Cherney DZI. Sotagliflozin and Kidney Outcomes, Kidney Function, and Albuminuria in Type 2 Diabetes and CKD: A Secondary Analysis of the SCORED Trial. Clin J Am Soc Nephrol. 2024 May 1;19(5):557-564. doi: 10.2215/CJN.0000000000000414. Epub 2024 Jan 26. PMID 38277468
- [Derived] Bhatt DL, Szarek M, Pitt B, Cannon CP, Leiter LA, McGuire DK, Lewis JB, Riddle MC, Inzucchi SE, Kosiborod MN, Cherney DZI, Dwyer JP, Scirica BM, Bailey CJ, Diaz R, Ray KK, Udell JA, Lopes RD, Lapuerta P, Steg PG; SCORED Investigators. Sotagliflozin in Patients with Diabetes and Chronic Kidney Disease. N Engl J Med. 2021 Jan 14;384(2):129-139. doi: 10.1056/NEJMoa2030186. Epub 2020 Nov 16. PMID 33200891
- [Derived] Cefalo CMA, Cinti F, Moffa S, Impronta F, Sorice GP, Mezza T, Pontecorvi A, Giaccari A. Sotagliflozin, the first dual SGLT inhibitor: current outlook and perspectives. Cardiovasc Diabetol. 2019 Feb 28;18(1):20. doi: 10.1186/s12933-019-0828-y. PMID 30819210

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 723 study centers in North America, Latin America, Western Europe, Eastern Europe, and the Rest of the World from 19 December 2017 to 08 July 2020.
Pre-assignment Details: Participants with a diagnosis of Type 2 diabetes (T2D), CV risk factors, and moderately impaired renal function were enrolled equally in 1 of 2 treatment groups, sotagliflozin or placebo.
Period: Overall Study
Arm/Group | Sotagliflozin | Placebo
Started | 5292 | 5292
Randomized and Treated | 5291 | 5286
Completed | 0 | 0
Not Completed | 5292 | 5292
Not completed — Death | 240 | 246
Not completed — Withdrawal by Subject | 57 | 68
Not completed — Site Terminated by Sponsor | 256 | 282
Not completed — Study Terminated by Sponsor | 4723 | 4664
Not completed — Reason not Specified | 16 | 32

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants analyzed according to the treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sotagliflozin | Placebo | Total
Number analyzed (Participants) | 5292 | 5292 | 10584
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.4) | 68.2 (8.4) | 68.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2347 | 2407 | 4754
  Male | 2945 | 2885 | 5830
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1671 | 1678 | 3349
  Not Hispanic or Latino | 3593 | 3581 | 7174
  Unknown or Not Reported | 28 | 33 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 205 | 216 | 421
  Asian | 317 | 365 | 682
  Native Hawaiian or Other Pacific Islander | 25 | 15 | 40
  Black or African American | 176 | 187 | 363
  White | 4383 | 4329 | 8712
  More than one race | 129 | 114 | 243
  Unknown or Not Reported | 57 | 66 | 123

OUTCOME MEASURES:

1. Primary Outcome: Number of Total Occurrences of Cardiovascular (CV) Death, Hospitalizations for Heart Failure (HHF) and Urgent Visits for Heart Failure (HF)
Description: Combined endpoint of the total number of occurrences (first and potentially subsequent) of CV death, HHF, and urgent HF visits after randomization. Events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 30 months
Population: ITT population included all randomized participants analyzed according to the treatment group allocated by randomization.
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 5292 | 5292
events per 100-person years | 5.6 | 7.5
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; The estimates of the hazard ratio (HR) and corresponding 2-sided 95% confidence interval (CI) was to be provided by a marginal Cox proportional hazard model stratified by region and ejection fraction, with non-cardiovascular (non-CV) death treated as a competing event; Test type: Superiority; p < 0.001, Cox proportional hazards model; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.63 to 0.88]

2. Secondary Outcome: Total Number of Occurrences of HHF and Urgent HF Visits
Description: Combined endpoint of the total occurrences (first and potentially subsequent) of HHF and urgent HF visits after randomization. Events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 30 months
Population: as for outcome 1
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 5292 | 5292
events per 100-person years | 3.5 | 5.1
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; The estimates of the HR and corresponding 2-sided 95% CI was to be provided by a marginal Cox proportional hazard model stratified by region and ejection fraction, with non-CV death treated as a competing event; Test type: Superiority; p < 0.001, Cox proportional hazards model; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.55 to 0.82]

3. Secondary Outcome: Number of Deaths From Cardiovascular Causes
Description: Number of events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 30 months
Population: as for outcome 1
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 5292 | 5292
events per 100-person years | 2.2 | 2.4
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.35, Cox proportional hazards model; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.73 to 1.12]

4. Secondary Outcome: Total Number of Occurrences of CV Death, HHF, Non-fatal Myocardial Infarction and Non-fatal Stroke
Description: Combined endpoint of the total number of occurrences (first and potentially subsequent) of CV death, HHF, non-fatal stroke, and non-fatal myocardial infarction after randomization. Events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 30 months
Population: as for outcome 1
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 5292 | 5292
events per 100-person years | 7.6 | 10.4
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.63 to 0.83]

5. Secondary Outcome: Total Number of Occurrences of HHF, Urgent HF Visit, CV Death, and HF While Hospitalized
Description: Combined endpoint of the total number of occurrences (first and potentially subsequent) after randomization of HHF, urgent HF visits, CV Death, and HF while hospitalized. Events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 30 months
Population: as for outcome 1
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 5292 | 5292
events per 100-person years | 6.4 | 8.3
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.65 to 0.89]

6. Secondary Outcome: Number of Occurrences After Randomization of the Composite of Sustained ≥50% Decrease in Estimated Glomerular Filtration Rate (eGFR) From Baseline (for ≥30 Days), Chronic Dialysis, Renal Transplant, or Sustained eGFR <15 mL/Min/1.73 m^2 (for ≥30 Days)
Description: Events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 30 months
Population: as for outcome 1
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 5292 | 5292
events per 100-person years | 0.5 | 0.7
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.46 to 1.08]

7. Secondary Outcome: Number of Deaths From Any Cause
Description: as for outcome 3
Time Frame: Up to 30 months
Population: as for outcome 1
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 5292 | 5292
events per 100-person years | 3.5 | 3.5
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; The estimates of the HR and corresponding 2-sided 95% CI was to be provided by a marginal Cox proportional hazard model stratified by region and ejection fraction; Test type: Superiority; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.83 to 1.18]

8. Secondary Outcome: Total Number of Occurrences of CV Death, Non-fatal Myocardial Infarction and Non-fatal Stroke
Description: Combined endpoint of the total number of occurrences (first and potentially subsequent) of CV death and urgent HF visits after randomization. Events that occurred during the study were calculated as the total number of events per 100 person-years of follow-up.
Time Frame: Up to 30 months
Population: as for outcome 1
Measure: Number; unit: events per 100-person years
Arm/Group | Sotagliflozin | Placebo
Number analyzed (Participants) | 5292 | 5292
events per 100-person years | 4.8 | 6.3
Statistical Analysis 1: Comparison: Sotagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.65 to 0.91]

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 10 days after the last dose of study drug (Up to 30 months)
Description: Number of Deaths (All causes) is based on all randomized participants (n=5292, 5292). Adverse Events are based on the Safety population that included all randomized participants who received at least 1 dose of investigational medicinal product (n=5291, 5286).
Arm/Group | Sotagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 246/5292 | 246/5292
Serious Adverse Events (participants affected / at risk) | 1236/5291 | 1331/5286
Other Adverse Events (participants affected / at risk) | 705/5291 | 609/5286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sotagliflozin (N=5291) | Placebo (N=5286)
Accelerated hypertension (Vascular disorders) | 0 | 2
Aortic dissection (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 1
Arterial haemorrhage (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 2
Deep vein thrombosis (Vascular disorders) | 6 | 15
Diabetic vascular disorder (Vascular disorders) | 3 | 0
Dry gangrene (Vascular disorders) | 6 | 4
Essential hypertension (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 8 | 13
Hypertensive crisis (Vascular disorders) | 7 | 13
Hypertensive emergency (Vascular disorders) | 4 | 1
Hypertensive urgency (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 5 | 7
Hypovolaemic shock (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 3 | 2
Internal haemorrhage (Vascular disorders) | 0 | 1
Leriche syndrome (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 2 | 1
Orthostatic hypotension (Vascular disorders) | 3 | 4
Pelvic venous thrombosis (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 16 | 15
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 4
Peripheral artery thrombosis (Vascular disorders) | 5 | 2
Peripheral embolism (Vascular disorders) | 1 | 1
Peripheral ischaemia (Vascular disorders) | 8 | 5
Peripheral vascular disorder (Vascular disorders) | 1 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 3
Subclavian steal syndrome (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 2 | 2
Varicose ulceration (Vascular disorders) | 0 | 1
Varicose vein (Vascular disorders) | 0 | 2
Vasculitis (Vascular disorders) | 1 | 0
Aortic aneurysm repair (Surgical and medical procedures) | 0 | 1
Aortic valve replacement (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 1
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Coronary angioplasty (Surgical and medical procedures) | 1 | 0
Foot amputation (Surgical and medical procedures) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 1 | 0
Intraocular lens implant (Surgical and medical procedures) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Knee operation (Surgical and medical procedures) | 0 | 1
Mitral valve replacement (Surgical and medical procedures) | 1 | 0
Nephrectomy (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 1 | 0
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bladder transitional cell carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Burkitt's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
External ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nasopharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour of the lung metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Oropharyngeal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary serous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 13
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Renal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 2
Asthenia (General disorders) | 2 | 2
Cardiac death (General disorders) | 3 | 0
Chest pain (General disorders) | 7 | 4
Chronic fatigue syndrome (General disorders) | 0 | 1
Death (General disorders) | 9 | 12
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 1
Influenza like illness (General disorders) | 0 | 1
Medical device site discharge (General disorders) | 0 | 1
Medical device site haematoma (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Necrobiosis (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 10 | 12
Oedema peripheral (General disorders) | 1 | 2
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 0
Soft tissue inflammation (General disorders) | 2 | 0
Sudden cardiac death (General disorders) | 14 | 8
Sudden death (General disorders) | 7 | 5
Systemic inflammatory response syndrome (General disorders) | 1 | 1
Vascular stent stenosis (General disorders) | 1 | 1
Acute stress disorder (Psychiatric disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 4 | 3
Conversion disorder (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Hallucination (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 7 | 4
Breast pain (Reproductive system and breast disorders) | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 2 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Testicular torsion (Reproductive system and breast disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Vulval disorder (Reproductive system and breast disorders) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Airway burns (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 7 | 7
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 2 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Colon injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 4 | 3
Dural tear (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 22 | 13
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 | 3
Femur fracture (Injury, poisoning and procedural complications) | 7 | 7
Fibula fracture (Injury, poisoning and procedural complications) | 4 | 2
Foot fracture (Injury, poisoning and procedural complications) | 12 | 15
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 7 | 4
Head injury (Injury, poisoning and procedural complications) | 7 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 5
Humerus fracture (Injury, poisoning and procedural complications) | 14 | 16
Incarcerated parastomal hernia (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1
Limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 4 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 4 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 2 | 4
Pelvic fracture (Injury, poisoning and procedural complications) | 3 | 0
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haematuria (Injury, poisoning and procedural complications) | 3 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Procedural shock (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 7 | 8
Rib fracture (Injury, poisoning and procedural complications) | 13 | 9
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 5
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Snake bite (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 4
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Stomal hernia (Injury, poisoning and procedural complications) | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 3 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 5 | 4
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haematoma (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 2 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 6 | 3
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 7 | 5
Alanine aminotransferase increased (Investigations) | 3 | 4
Blood bilirubin increased (Investigations) | 0 | 1
Blood glucose decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 5
Blood pressure increased (Investigations) | 1 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Catheterisation cardiac (Investigations) | 1 | 0
ECG signs of myocardial ischaemia (Investigations) | 1 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 1
Enterococcus test positive (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 2 | 3
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Klebsiella test positive (Investigations) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 3 | 1
Troponin increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 7 | 8
Acute left ventricular failure (Cardiac disorders) | 4 | 6
Acute myocardial infarction (Cardiac disorders) | 48 | 59
Acute right ventricular failure (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 18 | 25
Angina unstable (Cardiac disorders) | 44 | 52
Aortic valve sclerosis (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 3 | 3
Arrhythmia (Cardiac disorders) | 2 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 3
Atrial fibrillation (Cardiac disorders) | 34 | 35
Atrial flutter (Cardiac disorders) | 6 | 12
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 5 | 14
Atrioventricular block second degree (Cardiac disorders) | 5 | 3
Bifascicular block (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 7 | 7
Bundle branch block (Cardiac disorders) | 1 | 0
Cardiac aneurysm (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 5 | 11
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 94 | 147
Cardiac failure acute (Cardiac disorders) | 18 | 28
Cardiac failure chronic (Cardiac disorders) | 9 | 27
Cardiac failure congestive (Cardiac disorders) | 23 | 46
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 6 | 7
Cardiogenic shock (Cardiac disorders) | 6 | 5
Cardiohepatic syndrome (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 3
Coronary artery disease (Cardiac disorders) | 15 | 22
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery perforation (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 5 | 4
Heart valve incompetence (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 2 | 1
Left ventricular failure (Cardiac disorders) | 1 | 5
Microvascular coronary artery disease (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 24 | 55
Myocardial ischaemia (Cardiac disorders) | 6 | 7
Nodal arrhythmia (Cardiac disorders) | 1 | 1
Nodal rhythm (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 4 | 0
Prosthetic cardiac valve thrombosis (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 1
Sinus node dysfunction (Cardiac disorders) | 3 | 6
Subendocardial ischaemia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 2
Tachycardia (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 2
Ventricular extrasystoles (Cardiac disorders) | 2 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 4
Ventricular flutter (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 4 | 4
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 4
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 0 | 1
Blood loss anaemia (Blood and lymphatic system disorders) | 6 | 4
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 6 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 | 19
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Amnesia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Auditory nerve disorder (Nervous system disorders) | 0 | 1
Autonomic neuropathy (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 1
Brain injury (Nervous system disorders) | 1 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 4 | 2
Carpal tunnel syndrome (Nervous system disorders) | 2 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebellar stroke (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 4 | 6
Cerebral ischaemia (Nervous system disorders) | 1 | 4
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 13 | 16
Cerebrovascular disorder (Nervous system disorders) | 1 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 2
Cervicobrachial syndrome (Nervous system disorders) | 1 | 1
Dementia (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 2 | 0
Diabetic encephalopathy (Nervous system disorders) | 1 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 3 | 4
Disturbance in attention (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3
Dysarthria (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 2 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 8
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 1
Hemiparesis (Nervous system disorders) | 1 | 2
Hemiplegia (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 2
Hypoglycaemic coma (Nervous system disorders) | 1 | 1
Hypoglycaemic unconsciousness (Nervous system disorders) | 2 | 3
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 29 | 36
Lacunar infarction (Nervous system disorders) | 1 | 0
Lacunar stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 2 | 3
Lumbosacral radiculopathy (Nervous system disorders) | 2 | 3
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 2
Parkinsonism (Nervous system disorders) | 0 | 1
Post stroke seizure (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 3 | 1
Radiculopathy (Nervous system disorders) | 1 | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0
Sacral radiculopathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 5 | 1
Seizure (Nervous system disorders) | 2 | 2
Somnolence (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 26 | 27
Tension headache (Nervous system disorders) | 0 | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 6 | 14
Vascular encephalopathy (Nervous system disorders) | 1 | 0
Vertebral artery stenosis (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 2
Vertebrobasilar stroke (Nervous system disorders) | 1 | 0
Amaurosis fugax (Eye disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 5 | 5
Corneal degeneration (Eye disorders) | 0 | 1
Dermatochalasis (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 2 | 1
Diplopia (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1
Eyelid cyst (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 1
Macular fibrosis (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 2 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Retinal ischaemia (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 2
Vitreous haemorrhage (Eye disorders) | 2 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 6
Vertigo positional (Ear and labyrinth disorders) | 2 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 6
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 5
Diverticulum (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 | 2
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 5
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 3
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 2
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 3
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Mesenteric arterial occlusion (Gastrointestinal disorders) | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3
Obstructive pancreatitis (Gastrointestinal disorders) | 3 | 2
Oesophageal stent stenosis (Gastrointestinal disorders) | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 4
Pancreatitis acute (Gastrointestinal disorders) | 5 | 12
Pancreatitis chronic (Gastrointestinal disorders) | 4 | 3
Pancreatitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 2
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 4
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 2 | 6
Acute kidney injury (Renal and urinary disorders) | 61 | 52
Anuria (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 14 | 18
Cystitis glandularis (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 1
Diabetic end stage renal disease (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 3 | 4
Dysuria (Renal and urinary disorders) | 0 | 2
End stage renal disease (Renal and urinary disorders) | 0 | 1
Eosinophilic cystitis (Renal and urinary disorders) | 0 | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 0
Hydronephrosis (Renal and urinary disorders) | 3 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 8
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 2 | 5
Obstructive nephropathy (Renal and urinary disorders) | 0 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 2
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 2
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 11 | 16
Renal haematoma (Renal and urinary disorders) | 1 | 0
Renal hypertension (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 12 | 14
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Stag horn calculus (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 4
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 2 | 0
Ureterolithiasis (Renal and urinary disorders) | 4 | 3
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 4 | 5
Cholecystitis acute (Hepatobiliary disorders) | 10 | 10
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 5 | 4
Cholestasis (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0
Gallbladder rupture (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Pneumobilia (Hepatobiliary disorders) | 1 | 0
Device breakage (Product Issues) | 1 | 0
Device dislocation (Product Issues) | 0 | 1
Device failure (Product Issues) | 1 | 0
Device loosening (Product Issues) | 1 | 0
Device malfunction (Product Issues) | 0 | 1
Device occlusion (Product Issues) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 3
Cutaneous loxoscelism (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 14 | 9
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 0 | 1
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Oedema blister (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 3 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 12 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Crowned dens syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 | 12
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 1
Empty sella syndrome (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 0 | 1
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 5 | 9
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 17 | 25
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 11 | 4
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 | 6
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 23
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 14 | 11
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 35 | 31
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 9
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 2
Increased insulin requirement (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 14 | 1
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Metabolic syndrome (Metabolism and nutrition disorders) | 2 | 2
Obesity (Metabolism and nutrition disorders) | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1
Abdominal abscess (Infections and infestations) | 2 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 5 | 5
Abscess neck (Infections and infestations) | 0 | 1
Acarodermatitis (Infections and infestations) | 1 | 0
Acute endocarditis (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 4 | 3
Arthritis bacterial (Infections and infestations) | 1 | 4
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 3
Bacterial colitis (Infections and infestations) | 0 | 1
Bacterial parotitis (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 2
Bacterial sepsis (Infections and infestations) | 4 | 2
Bronchitis (Infections and infestations) | 0 | 7
Bronchitis bacterial (Infections and infestations) | 2 | 5
Bronchitis viral (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 5 | 6
COVID-19 pneumonia (Infections and infestations) | 6 | 5
Campylobacter colitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 22 | 17
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 2 | 0
Cholecystitis infective (Infections and infestations) | 0 | 1
Chronic hepatitis B (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 3 | 2
Cryptosporidiosis infection (Infections and infestations) | 1 | 0
Cutaneous leishmaniasis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 6 | 3
Cystitis bacterial (Infections and infestations) | 7 | 8
Cystitis escherichia (Infections and infestations) | 1 | 3
Cystitis klebsiella (Infections and infestations) | 1 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 1
Dengue haemorrhagic fever (Infections and infestations) | 0 | 1
Dermo-hypodermitis (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 9 | 4
Diabetic gangrene (Infections and infestations) | 4 | 0
Diverticulitis (Infections and infestations) | 5 | 2
Dysentery (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 2
Erysipelas (Infections and infestations) | 6 | 10
Escherichia infection (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 3 | 3
Fournier's gangrene (Infections and infestations) | 1 | 2
Fungaemia (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 3 | 8
Gastroenteritis (Infections and infestations) | 18 | 10
Gastroenteritis bacterial (Infections and infestations) | 0 | 1
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 5 | 1
Genital abscess (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 1
Groin infection (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 2 | 3
Impetigo (Infections and infestations) | 0 | 1
Infected cyst (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 2 | 4
Infection (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 3 | 7
Injection site abscess (Infections and infestations) | 1 | 0
Intestinal fistula infection (Infections and infestations) | 0 | 1
Keratitis bacterial (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 1
Liver abscess (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 3
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 2
Lower respiratory tract infection viral (Infections and infestations) | 1 | 1
Ludwig angina (Infections and infestations) | 1 | 0
Mastitis bacterial (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0
Medical device site infection (Infections and infestations) | 0 | 1
Meningoencephalitis bacterial (Infections and infestations) | 1 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0
Myocarditis infectious (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 2
Nephritis bacterial (Infections and infestations) | 0 | 1
Ophthalmic herpes simplex (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 3 | 0
Osteomyelitis (Infections and infestations) | 9 | 8
Osteomyelitis acute (Infections and infestations) | 2 | 2
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Otitis media bacterial (Infections and infestations) | 1 | 0
Ovarian abscess (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Peptic ulcer helicobacter (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 4 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Periumbilical abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 37 | 57
Pneumonia adenoviral (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 17 | 39
Pneumonia haemophilus (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 3 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 2
Pneumonia viral (Infections and infestations) | 3 | 2
Post procedural pneumonia (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 6 | 1
Psoas abscess (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 3 | 2
Pulmonary tuberculosis (Infections and infestations) | 1 | 1
Pyelitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 10 | 10
Pyelonephritis acute (Infections and infestations) | 7 | 4
Pyelonephritis chronic (Infections and infestations) | 3 | 3
Q fever (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 13 | 12
Septic shock (Infections and infestations) | 3 | 4
Sinusitis aspergillus (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 2 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 4 | 1
Subdiaphragmatic abscess (Infections and infestations) | 0 | 1
Suspected COVID-19 (Infections and infestations) | 1 | 0
Systemic infection (Infections and infestations) | 1 | 0
Systemic viral infection (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 8 | 10
Urinary tract infection bacterial (Infections and infestations) | 9 | 13
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 12 | 10
Vestibular neuronitis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 2 | 1
Viral myocarditis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Vulval cellulitis (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sotagliflozin (N=5291) | Placebo (N=5286)
Diarrhoea (Gastrointestinal disorders) | 373 | 253
Hypoglycaemia (Metabolism and nutrition disorders) | 380 | 395

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to business decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must provide any proposed publication or presentation to Sponsor for Sponsor's review, comment and approval at least thirty (30) days prior to the proposed submission for publication date or the proposed presentation date. Sponsor shall have the right to have deleted from the final version of the publication any confidential information, proprietary information, or patentable subject matter.

DOCUMENTS (2):
  • Study Protocol (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT03315143/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT03315143/SAP_001.pdf